CLINICAL TRIAL: NCT06130618
Title: The Effects of Ultrasound Guided Ozone and Lidocaine Injections on Pain, Functional Level and Posture in Piriformis Syndrome
Brief Title: The Effects of Ultrasound Guided Ozone and Lidocaine Injections in Piriformis Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Bilge Kesikburun, Associate Professor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2-23-4633
Record Dates: First submitted 2023-11-03; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Piriformis Syndrome
MeSH Terms: conditions — Piriformis Muscle Syndrome | interventions — Ozone; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozone injection (Active Comparator): After localizing the piriformis muscle with ultrasound guidance, 5 ml - 20 μg/mL ozone will be injected.
  Interventions: Other: Ozone
- Lidocaine injection (Active Comparator): After localizing the piriformis muscle with ultrasound guidance, 5 ml - 2% lidocaine will be injected.
  Interventions: Drug: Lidocain

INTERVENTIONS:
Other: Ozone — After localizing the piriformis muscle and sciatic nerve with ultrasound guidance, 5 ml - 20 μg/mL ozone will be injected.
  Other Names: Ozone injection
  Arms: Ozone injection
Drug: Lidocain — After localizing the piriformis muscle and sciatic nerve with ultrasound guidance, 5 ml - 2% lidocaine will be injected.
  Other Names: Lidocaine injection
  Arms: Lidocaine injection

SUMMARY:
Piriformis Syndrome (PS) is defined as a trap neuropathy that involves compression of the sciatic nerve by the piriformis muscle, leading to a number of symptoms along with sciatic pain, initially in the hip muscles. In clinical practice, it is estimated to be between 12.2-27%.

Repetitive movements with increased demand on the piriformis muscle can lead to increased muscle tension, compression of the sciatic nerve within the muscle, and the development of PS. Additionally, the anatomical structure of the piriformis muscle and the alignment and damage of adjacent structures play a role in the pathophysiology of sciatic nerve compression in PS. It is considered in pathophysiology that a morphological change (contracture, hypertrophy) may cause compression of the sciatic nerve or the relationships of different anatomical structures that change with biomechanical restrictions.

Pain is observed along the ipsilateral sciatic nerve distribution due to compression of the sciatic nerve. Additionally, it has been observed that patients with PS are accompanied by weakness in the gluteal muscles, mostly in the gluteus maximus and medius muscles. Accompanying weakness has an effect on static and dynamic posture (2,3). The negative effect of pain on posture has also been shown in studies (4). Pain and muscle changes in the lower extremities also cause disability and postural instability. It has been reported that static and dynamic postural balance is reduced in PS compared to healthy controls (1).

Conservative treatment for PS significantly reduces pain with a wide range of therapeutic alternatives. Since ozone injection does not have side effects or major complications, its use in the treatment of myofascial pain syndromes and piriformis syndrome is supported by studies (5). It has an analgesic effect, increasing the pain threshold by activating serotonin-mediated pathways to release endogenous opioids. Additionally, it is used safely due to its low side effect profile. In the literature, it has been shown that local anesthetic injection applications alone or in combination with steroids are effective in the treatment of PS alone due to the therapeutic effects of local anesthetic (6).

This study aimed to investigate the effects of ozone and local anesthetic injection on pain, functional level and posture in patients diagnosed with PS.

DETAILED DESCRIPTION:
It was planned as a randomized controlled study. Patients diagnosed with Priformis Syndrome will be evaluated and their demographic data and examination information will be recorded.

Patients will be divided into 2 groups: ozone and lidocaine injections by computerized randomization. If there is a contraindication for ozone, the patient will be included in the lidocaine group, and similarly, if the patient has a contraindication for lidocaine, the patient will be included in the ozone group. According to G-power analysis, a total of 28 patients, 14 for each group, will be included in the study.

One group will be injected with 5 mL of lidocaine 2% after localizing the piriformis muscle with USG guidance, and the other group will be injected with 5 ml - 20 μg/mL ozone after localizing the piriformis muscle with USG guidance.

Pain levels of the patients will be evaluated with the visual analog scale at baseline, 1st Week, 1st Month and 3rd Month. Functional levels of all patients will be measured using the Lower Extremity Functional Scale; Posture evaluation includes trunk imbalance (sagittal/coronal imbalance), vertebral rotation, apical deviation, pelvic tilt, pelvic torsion, pelvic obliquity, kyphotic angle, lordotic angle measurement with DIERS 4D posture analyzer, static balance parameters with HUR balance device will be evaluated at baseline and at the 3rd month.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients with pain in the posterior aspect of the thigh and diagnosed with piriformis through physical examination and special tests
* Knowing how to read and write Turkish
* Patients with visual analog scale ≥5

Exclusion Criteria:

* Those with a history of lumbar discopathy or a history of discopathy surgery
* BMI over ≥ 30
* Having had a corticosteroid injection within the last 3 months
* Presence of neurological deficit in the lower extremity
* Having a history of previous hip surgery
* Having progressive or non-progressive central and peripheral nervous system disease,
* Patients in pregnancy and lactation
* Use of anticoagulants

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain condition will evaluate by the visual analog scale | Baseline, 1. week, 1. month, 3. month
  The Visual Analog Scale (VAS) pain score (on a range of 0-10, with 0 representing no pain and 10 representing the severe pain) will evaluate.
posture | Baseline, 3. month
  Posture Analysis will be evaluated by DIERS formetric 4D. Participants will be positioned two meters away from the camera unit and formetric 4D projection. The device will project light stripes on the back of the participant. The back's surface will be captured on camera, converted to digital data, and displayed in three dimensions. Every scan will record 12-13 images over 6 seconds (2 Hz), and the manufacturer's recommendations will be followed for processing. Spinal reference points, measures of the spinal curve, distance and localization, imbalances of the trunk and pelvis, and spinal deviation will be measured. Spine shape parameters are expressed in millimeters, percentages, or degrees depending on the specific parameter.
Balance | Baseline, 3. month
  The static and dynamic postural control were measured by the HUR SmartBalance BTG4 system (Hur Labs, Tampere, Finland). Participants were asked to stand barefoot on the balance platform, and were requested to stand as quietly as possible, without moving and looking forward, during the measurement. The stable floor was the platform's own floor, while the unstable floor was the foam cushion given by the manufacturer with the device. Data were collected for 30 seconds. The following parameters were calculated from the center of pressure (CoP) displacement time series for static postural control: sway area, trace length, velocity, Romberg, lateral sway, anterior-posterior sway. The limits of stability (LOS) were used to determine the dynamic postural control. The patients were asked to tilt their bodies forward, backward, leftward, and rightward for 8 seconds in each direction.

SECONDARY OUTCOMES:
Function | Baseline, 3. month
  The Lower Extremity Functional Scale (LEFS) is a set of 20 questions designed to assess an individual's capacity to carry out routine tasks. The highest possible score is 80. The lower the score means the higher the disability.

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Kesikburun, Ass. Prof, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
When the study is completed study protocol and Clinical Study Report will be shared.
Supporting Information: Study Protocol, CSR
Time Frame: When the study is completed
Access Criteria: Data will be shared in case of reasonable request.

REFERENCES:
- [Background] Jardak M, Chaari F, Bouchaala F, Fendri T, Harrabi MA, Rebai H, Sahli S. Does piriformis muscle syndrome impair postural balance? A case control study. Somatosens Mot Res. 2021 Dec;38(4):315-321. doi: 10.1080/08990220.2021.1973404. Epub 2021 Sep 14. PMID 34519264
- [Background] Chon J, Kim HS, Lee JH, Yoo SD, Yun DH, Kim DH, Lee SA, Han YJ, Soh Y, Kim Y, Han YR, Won CW, Han S. Association Between Asymmetry in Knee Extension Strength and Balance in a Community-Dwelling Elderly Population: A Cross-Sectional Analysis. Ann Rehabil Med. 2018 Feb;42(1):113-119. doi: 10.5535/arm.2018.42.1.113. Epub 2018 Feb 28. PMID 29560331
- [Background] Bouche K, Stevens V, Cambier D, Caemaert J, Danneels L. Comparison of postural control in unilateral stance between healthy controls and lumbar discectomy patients with and without pain. Eur Spine J. 2006 Apr;15(4):423-32. doi: 10.1007/s00586-005-1013-4. Epub 2005 Aug 18. PMID 16133081
- [Background] Misirlioglu TO, Akgun K, Palamar D, Erden MG, Erbilir T. Piriformis syndrome: comparison of the effectiveness of local anesthetic and corticosteroid injections: a double-blinded, randomized controlled study. Pain Physician. 2015 Mar-Apr;18(2):163-71. PMID 25794202